CLINICAL TRIAL: NCT01048164
Title: Measuring the Effect of Therapeutic Massage on Pain and Discomfort in Cardiac Cath Lab Staff - A Pilot Study
Brief Title: Measuring the Effect of Therapeutic Massage on Pain and Discomfort in Cardiac Cath Lab Staff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Deborah Engen, OT, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 08-000190
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Stress; Fatigue; Anxiety
Keywords: Massage; Relaxation
MeSH Terms: conditions — Fatigue; Anxiety Disorders | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 10 Massages (Active Comparator): This group consists of individuals that wear lead aprons, and they will receive ten, 30-minute scheduled massage appointments during the hours the participant is working in the cardiac lab, over a 10 week period.
  Interventions: Procedure: Massage
- 5 Massages (Active Comparator): This group consists of individuals that wear lead aprons, and they will receive five, 30-minute scheduled massage appointments, during the hours the participant is working in the cardiac lab, over a 5 week period. This arm will not receive massages for the first 5 weeks and then will receive their massages during the second 5 week period.
  Interventions: Procedure: Massage
- Control Group (No Intervention): This group will consist of those individuals that wear lead aprons with no desire to participate in the massage study yet are willing to provide information through questionnaires. They will be given the same questionnaire as those in the two massage therapy arms of the study, at the beginning, middle, and end of study.

INTERVENTIONS:
Procedure: Massage — Chair Massage
  Arms: 10 Massages; 5 Massages

SUMMARY:
The purpose of this study is to evaluate the effect of therapeutic massage in alleviating musculoskeletal pain and discomfort associated with wearing lead aprons in the cardiac cath lab. We also want to evaluate if therapeutic massage will reduce fatigue, stress, and anxiety while improving the level of relaxation in cardiac cath lab employees who wear lead aprons.

DETAILED DESCRIPTION:
The cardiac catheterization laboratory is a very dynamic work environment. The physical and psychosocial demands of the work environment place a significant amount of stress on the physical well being of the employee. The nature of the work involved includes that of responding to rapidly changing patient clinical conditions which are often urgent, and require repetitive actions in an ergonomically challenging environment. In addition, employees who are directly exposed to the radiation required to perform diagnostic and interventional procedures wear lead aprons weighing on average 10-15 pounds.

A constant build-up of tension in the muscles from regular, repetitive activity may lead to stresses on the muscles, joints, ligaments and tendons. Adding to this, working while wearing lead aprons, with elements of repetitive use and non-optimal ergonomic situations, Cardiac Cath Lab employees are at higher risk for muscle imbalances. The accumulation of tension and imbalance leads to joint wearing and muscle fatigue that result in injuries. Massage therapy, applied skillfully, is one of the most effective forms of therapy for releasing muscle tension, restoring balance to the musculoskeletal system, while creating awareness of musculoskeletal balance in the employee. Massage provided regularly may help employees prevent injuries caused by overuse.

As muscle imbalances develop they often go undiagnosed until they are serious enough to cause the employee discomfort or impede performance. Frequently the discomfort is masked with pain medications and ultimately leads to injuries. A skilled massage therapist will detect variations in the soft tissues and by using the correct techniques, help the employee maintain a much healthier physical state and prevent injury.

Massage therapy is purported to affect both the structure and function of the musculoskeletal system by promoting the relaxation response and reducing muscle tension and fatigue while improving posture. Given the potential benefits of massage therapy, many work environments are implementing massage therapy programs to improve the health and well being of their employees.

ELIGIBILITY:
Inclusion Criteria:

Diagnostic and interventional cardiology staff including:

* cardiologists
* cardiology fellows
* nurses
* technical staff
* and a core group of CRNA's employed by the Cardiac Catheterization Laboratory.

These staff members, per their job descriptions, wear lead aprons while caring for patients during the weeks of the massage therapy pilot study.

Exclusion Criteria:

* Individuals that decline to participate in the study.
* Massage therapy has contraindications that require a physician's order before the therapist is allowed to see the person for massage. The following total contraindications will be total exclusions for this study unless the individual gains a physician's order that negates the exclusions or defines it to a local contraindication.

Total Contraindications

* Acute sprain with swelling
* Lymphatic cancer
* Fever

Local Contraindications do not exclude the person from the study. These are area exclusions that disallow the therapist to work on a specific part of the body and/or the therapist needs to adjust techniques. The therapist will track all local contraindications.

Local contraindications:

* Varicose veins
* Pregnancy
* Trapped or pinched nerve (radicular symptoms)
* Skin abrasions, open wounds
* Venous thrombus
* Melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Compare and contrast the level of pain and discomfort in staff that wear lead aprons at baseline, end of first 5-weeks of massage therapy, end of the second 5-weeks of massage therapy and to those that do not get massage during that same period. | 10 Weeks

SECONDARY OUTCOMES:
Compare the level of stress, anxiety, and relaxation in staff that wear lead aprons, at baseline, end of first 5-weeks of massage therapy, end of the second 5-weeks of massage therapy and to those that do not get massage during that same period. | 10 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shelly R. Keller, R.N., C.N.P., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Keller SR, Engen DJ, Bauer BA, Holmes DR Jr, Rihal CS, Lennon RJ, Loehrer LL, Wahner-Roedler DL. Feasibility and effectiveness of massage therapy for symptom relief in cardiac catheter laboratory staff: a pilot study. Complement Ther Clin Pract. 2012 Feb;18(1):4-9. doi: 10.1016/j.ctcp.2011.08.006. Epub 2011 Sep 23. PMID 22196566